CLINICAL TRIAL: NCT04978324
Title: Scaling and Root Planning With Localized Delivery of Autogenous Growth Factors- Platelet Rich Fibrin (PRF): A Randomized Split-mouth Clinical Trial
Brief Title: Scaling and Root Planning With Localized Delivery of Autogenous Growth Factors- Platelet Rich Fibrin (PRF)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Fellow graduated before successfully enrolling any participants
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20021781
Record Dates: First submitted 2021-07-16; First posted 2021-07-27 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Periodontitis Chronic Generalized Severe; Periodontitis Chronic Generalized Moderate
MeSH Terms: interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autogenous Growth Factors Left Side (Experimental): 5-8mm pockets on the left side of the mouth will receive insertion of small treatment after deep cleaning. The right side of the mouth will receive deep cleaning only, the standard of care.
  Interventions: Biological: leukocyte platelet rich fibrin (L-PRF); Procedure: Scaling and Root Planing
- Autogenous Growth Factors Right Side (Experimental): 5-8mm pockets on the right side of the mouth will receive insertion of small treatment after deep cleaning. The left side of the mouth will receive deep cleaning only, the standard of care.
  Interventions: Biological: leukocyte platelet rich fibrin (L-PRF); Procedure: Scaling and Root Planing

INTERVENTIONS:
Biological: leukocyte platelet rich fibrin (L-PRF) — Participants blood will be spun to obtain L-PRF strips and liquid L-PRF. Pockets will receive insertion of small L-PRF strips followed by liquid L-PRF injections to fill the 5-8mm pockets of the test side.
Procedure: Scaling and Root Planing — Scaling and root planing, which is the standard of care, will be performed on the control side using Cavitron and hand scalers on test and control sides under local anesthesia.

SUMMARY:
The purpose of this research study is to find out about the effect of growth factors extracted from blood on improving healing of periodontal pockets (Gum pockets) after deep gum cleaning.

DETAILED DESCRIPTION:
Blood has a lot of cells that help with healing and regeneration. These cells could be obtained by spinning blood in a centrifuge machine which allows the cells to separate at high spinning forces. After spinning, the blood will be separated into 3 different layers. The middle layer has the highest concentration of cells that help in healing and it is called the leukocyte platelet rich plasma (L-PRF).

The aim of this study is to use participant's own blood to retrieve (L-PRF) and place it in the diseased tissue around teeth, after the deep cleaning, to examine its effect in improving the healing and compare the results with gum pockets that haven't received L-PRF

In this study, participants will be asked to do the following things:

1. Visit VCU Graduate Periodontics clinic 6 times for scheduled study visits after the initial periodontal exam.:

   * 1st appointment: A digital impression of upper and lower teeth using an intraoral scanner, a light source laser that will capture digital impressions of the teeth, will be taken. These digital impressions will be used to create removable resin stents that fit on top of the teeth which will help in obtaining accurate and reproducible clinical measurements. The stents will be used on almost all participant's visits to the graduate periodontics clinic for the duration of the study for data collection.
   * 2nd and 3rd appointment: The deep cleaning will be divided into 2 appointments which should be less than 2 weeks apart. During each appointment, one arch, either the upper or the lower arch, will be scaled and root planed. Local anesthesia will be used to anesthetize the participant before the cleaning. Ultrasonic cleaner and hand instruments will be used for the deep cleaning. After finishing the deep cleaning, 36 ml of participant's blood will be collected in 4 tubes through the antecubital vein. The tubes will be spun in an FDA approved spinning machine to obtain the liquid and membrane forms of the L-PRF. The L-PRF will then be inserted in the test sites on one side of the arch while the other side will not receive the L-PRF.
   * 4th appointment: Prophylaxis and plaque control 2 weeks after 2nd appointment.
   * 5th appointment: Evaluation of deep periodontal cleaning and data collection 4-5 weeks after the 2nd appointment
   * 6th appointment: Periodontal cleaning and data collection 3 months after 2nd appointment.
2. Follow the oral hygiene instructions given

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (ASA 1 or 2) adults over the age of 18
* A similar number of bilateral 5-8 mm pocket depths
* Diagnosed with Stage II or Stage III chronic periodontitis.

Exclusion Criteria:

* Uncontrolled systemic illness that may affect healing or clotting such as diabetes mellitus, immunocompromisation, bleeding disorders, ongoing chemo- or radiotherapy
* Active smokers
* Pregnancy
* Periodontal treatment in the last six months
* Antibiotic therapy within three months prior to treatment
* Taking medications that could affect periodontal status or healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in probing depths (PD) | Baseline to 6 months
  PD will be measured from the gingival margin to pocket base using a participant specific fabricated removable resin stent with an assigned #15 UNC probe.
Change in clinical attachment level (CAL) | Baseline to 6 months
  CAL will be measured from cemento-enamel junction CEJ to the base of the pocket using the same stent as PD
Bleeding on probing (BOP) | Baseline to 6 months
  Bleeding on probing (BOP) will be recorded on an ordinal scale where sites that will bleed on probing will be given a score of 1 while sites that don't bleed will be given a score of 0.
Plaque index (PI) | Baseline to 6 months
  PI will be recorded using the Loe and Silness Index. Scores range from 0 - No plaque to 3 - Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Gingival index | Baseline to 6 months
  GI will be recorded using the Loe and Silness gingival index. Scores range from 0 - Normal gingiva to 3 - Severe inflammation - marked redness and edema, ulceration. Tendency toward spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Waldrop, DDS, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No